CLINICAL TRIAL: NCT00885079
Title: Confirmatory Study of OPC-12759 Ophthalmic Suspension in Dry Eye Patients
Brief Title: Confirmatory Study of OPC-12759 Ophthalmic Suspension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 037E-08-001
Record Dates: First submitted 2009-04-19; First posted 2009-04-21 (Estimated); Results first posted 2013-12-12 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-11

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rebamipide (Experimental): Instillation,4 times/day for 4 weeks
  Interventions: Drug: OPC-12759 Ophthalmic suspension
- Hyaluronate (Active Comparator): Instillation,6 times/day for 4 weeks
  Interventions: Drug: Hyalein Mini Ophthalmic solution

INTERVENTIONS:
Drug: OPC-12759 Ophthalmic suspension — OPC-12759 Ophthalmic suspension 2%
  Arms: Rebamipide
Drug: Hyalein Mini Ophthalmic solution — Hyalein Mini Ophthalmic solution 0.1%
  Arms: Hyaluronate

SUMMARY:
The purpose of this study is to verify whether OPC-12759 ophthalmic suspension is effective compared with active control in dry eye patients.

ELIGIBILITY:
Inclusion Criteria:

1. Out patient
2. Subjective complaint of dry eye that has been present for minimum 20 months
3. Ocular discomfort severity is moderate to severe
4. Corneal - conjunctival damage is moderate to severe
5. Unanesthetized Schirmer's test score of 5mm/5minutes or less
6. Best corrected visual acuity of 0.2 or better in both eyes

Exclusion Criteria:

1. Presence of anterior segment disease or disorder other than that associated with keratoconjunctivitis sicca
2. Ocular hypertension patient or glaucoma patient with ophthalmic solution
3. Anticipated use of any topically-instilled ocular medications or patients who cannot discontinue the use during the study
4. Anticipated use of contact lens during the study
5. Patient with punctal plug
6. Any history of ocular surgery within 12 months
7. Female patients who are pregnant,possibly pregnant or breast feeding
8. Known hypersensitivity to any component of the study drug or procedural medications
9. Receipt of any investigational product within 4 months.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2009-05; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eiji Murakami, Study Chair — OPCJ-DDO
Locations (5):
- Japan (5):
  - Kyushu region, Kagoshima
  - Chushikoku region, Matsuyama
  - Tokai region, Nagoya
  - Kansai region, Osaka
  - Kanto region, Tokyo

RESULTS

PARTICIPANT FLOW:
Groups:
- Rebamipide: Instillation,4 times/day for 4 weeks
  OPC-12759 Ophthalmic suspension : OPC-12759 Ophthalmic suspension 2%
- Hyaluronate: Instillation,6 times/day for 4 weeks
  Hyalein Mini Ophthalmic solution : Hyalein Mini Ophthalmic solution 0.1%
Period: Overall Study
Arm/Group | Rebamipide | Hyaluronate
Started | 93 | 95
Completed | 91 | 91
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rebamipide | Hyaluronate | Total
Number analyzed (Participants) | 93 | 95 | 188
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 55 | 59 | 114
  >=65 years | 38 | 36 | 74
Age Continuous [Mean (Standard Deviation); unit: years] | 58.0 (17.7) | 55.2 (16.9) | 56.6 (17.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 80 | 163
  Male | 10 | 15 | 25
Region of Enrollment [Number; unit: participants]
  Japan | 93 | 95 | 188

OUTCOME MEASURES:

1. Primary Outcome: Change in Fluorescein Corneal Staining (FCS) Score From Baseline
Description: FCS indicates the damage to the corneal epithelium. Per the National Eye Institute/Industry Workshop report, the cornea was divided into 5 fractions, each of which was given a staining score from 0 to 3, and the total score was calculated (0-15). 0 is better. Noninferiority for change from baseline in the FCS score (LOCF) was determined by comparing the noninferiority margin (0.4) with the upper limit of the 95% confidence interval (CI) of the difference between the 2 treatment groups
Time Frame: Baseline, Weeks4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rebamipide | Hyaluronate
Number analyzed (Participants) | 93 | 95
units on a scale | -3.7 (0.3) | -2.9 (0.2)
Statistical Analysis 1: Comparison: Rebamipide vs Hyaluronate; Test type: Non-Inferiority or Equivalence — Non-inferiority for change from baseline in the FCS score was determined by comparing the non-inferiority margin (0.4) with the upper limit of the confidence interval of the difference between the 2 treatment groups; p < 0.05, t-test, 2 sided — An analysis of change from baseline of FCS was performed using t-test. The level of singnificanse was 5 % (2-sided); Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-1.47 to -0.24], Standard Deviation 2.1

2. Primary Outcome: Change in Lissamine Green Conjunctival Staining (LGCS) Score From Baseline
Description: LGCS indicates the damage to the conjunctival epithelium. Per the National Eye Institute/Industry Workshop report, the conjunctiva was divided into 6 fractions, each of which was given a staining sdore from 0 to 3, and the total score was calculated (0-18). 0 is better. Superiority was verified by comparing t-test results for change from baseline in the LGCS score (LOCF) between 2 treatment groups.
Time Frame: Baseline, Weeks4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rebamipide | Hyaluronate
Number analyzed (Participants) | 93 | 95
units on a scale | -4.5 (3.2) | -2.4 (2.5)
Statistical Analysis 1: Comparison: Rebamipide vs Hyaluronate; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = -2.1

ADVERSE EVENTS:
Arm/Group | Rebamipide | Hyaluronate
Serious Adverse Events (participants affected / at risk) | 0/93 | 0/95
Other Adverse Events (participants affected / at risk) | 27/93 | 19/95
OTHER ADVERSE EVENTS (reported when occurring in more than 1.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rebamipide (N=93) | Hyaluronate (N=95)
Blepharitis (Eye disorders) | 0 (0) | 1 (1)
Chalazion (Eye disorders) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 2 (2)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Erythema of eyelid (Eye disorders) | 0 (0) | 1 (1)
Eye discharge (Eye disorders) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 2 (2)
Eye pain (Eye disorders) | 0 (0) | 3 (3)
Eyelid oedema (Eye disorders) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 2 (2) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 1 (1) | 1 (1)
Eye pruritus (Eye disorders) | 4 (4) | 2 (2)
Ocular discomfort (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Thirst (General disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Foreign body in eye (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1)
Blood potassium increased (Investigations) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 1 (1)
Blood urine present (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 3 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (bitter taste) (Nervous system disorders) | 9 (9) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No